CLINICAL TRIAL: NCT05534672
Title: Multicenter, Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy and Safety of Rapamycin in Drug Resistant Epilepsy Associated With TSC
Brief Title: Placebo Controlled Study to Assess the Efficacy and Safety of Rapamycin in Drug Resistant Epilepsy Associated With Tuberous Sclerosis Complex
Acronym: RaRE-TS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Katarzyna Kotulska (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Kotulska, Head of the Department of Neurology and Epileptology at The Children's Memorial Health Institute, Children's Memorial Health Institute, Poland
Organization: Children's Memorial Health Institute, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RaRE-TS
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Tuberous Sclerosis Complex
Keywords: tuberous sclerosis complex, epilepsy, rapamycin, drug resistant epilepsy
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy; Drug Resistant Epilepsy | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapamycin arm (Experimental): Each patient randomized to the rapamycin arm will receive rapamycin in liquid. The rapamycin will be administered in individually calculated doses depending on the body surface of participants
  Interventions: Other: Rapamycin
- Placebo arm (Placebo Comparator): The patients assigned to the placebo arm will receive placebo in liquid, analogically to the rapamycin group.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Rapamycin — Rapamycin in liquid administered orally
  Arms: Rapamycin arm
Other: Placebo — Placebo in liquid administered orally
  Arms: Placebo arm

SUMMARY:
The purpose of the RaRE-TS study is to determine safety, tolerability and efficacy of rapamycin versus placebo in a drug resistant epilepsy associated with tuberous sclerosis complex (TSC).

DETAILED DESCRIPTION:
This is a two-arm, randomized, double-blind, placebo controlled study to evaluate the efficacy, tolerability, and safety of rapamycin versus placebo in a drug resistant epilepsy associated with TSC. The study consists of 3 phases for each patient: screening, dose adjustment blinded phase, core blinded phase, followed by open-label observation. Patients who meet the eligibility criteria will be randomized to receive rapamycin or placebo. The randomization ratio is 1:1. Randomization will be stratified by age, sex and and the number of antiepileptic drugs ever used in the patient's history (up to 3 drugs / more than 3 drugs).

ELIGIBILITY:
Inclusion Criteria:

* male or female aged from 3 months up to 50 years at the day of randomization
* patients/parents/caregivers are willing to and able to give informed consent form for the participation in the study
* patients/parents/caregivers are willing to and able to comply with all study requirements
* definite diagnosis of TSC according to the Consensus criteria (Northrup, 2013)
* drug-resistant epilepsy associated with TSC with at least 8 seizures during 4 weeks

Exclusion Criteria:

* history of treatment with mTOR inhibitor in the three months prior to screening,
* history of pseudo-epileptic seizures,
* history of progressive CNS disease other than TSC
* recent surgery within 2 weeks prior to the screening
* severe infection within 2 weeks prior to the screening
* use of the cannabis derivatives
* contraindications for MRI or general anesthesia
* occurrence of the serious comorbidities which, in the opinion of the investigator, may either put a patient at significant risk associated with the participation in the study or may influence the results of the study the investigator
* pregnancy

Ages: 3 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
comparison of the number of patients with at least 50% reduction of seizures per week in the last month of the core blinded phase in comparison to screening phase in the rapamycin vs placebo group | final analyses after the formal final database lock, planned within one month after the last patient last visit in the study
number of adverse events (according to CTCAE classification) in the rapamycin vs placebo group during the double-blind core phase | final analyses after the formal final database lock, planned within one month after the last patient last visit in the study

SECONDARY OUTCOMES:
comparison of the number of seizures per week and the number of days free of seizures in the rapamycin vs placebo group, during 12-week treatment in double-blind core phase | final analyses after the formal final database lock, planned within one month after the last patient last visit in the study
severity of adverse events (according to CTCAE) and the number of patients withdrawn from the study due to adverse events in the rapamycin vs placebo group | final analyses after the formal final database lock, planned within one month after the last patient last visit in the study

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Medical University of Lodz, Lodz
  - Children's Memorial Health Institute, Neurology and Epileptology, Warsaw